CLINICAL TRIAL: NCT06932354
Title: Metabolic Monitoring During Therapeutic Hypothermia (Cooling) for Hypoxic Ischaemic Encephalopathy
Acronym: MeCool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathryn Beardsall (Other)
Responsible Party: Sponsor-Investigator, Kathryn Beardsall, Principle Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 251956
Record Dates: First submitted 2021-01-26; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CGM — masked continuous glucose monitoring

SUMMARY:
This study aims to determine if CGM can be safely used in these babies, and to use this alongside innovative methods to measure alternative fuels to optimise care of these vulnerable babies.

DETAILED DESCRIPTION:
In the UK approximately 1200 babies per year undergo 'cooling' for the treatment of 'birth asphyxia' or hypoxic ischaemic encephalopathy (HIE). HIE not only impacts on brain metabolism but disturbs the normal metabolic balance in these babies who are at risk of hypoglycaemia and hyperglycaemia, which may exacerbate the effect of their primary brain injury. The clinical significance of hypoglycaemia is dependent on the availability of alternative fuels such as ketones and lactate. Clinical management of glucose control in these extremely ill babies is challenging because of infrequent blood glucose measurements and inability to measure alternative fuels. We have used continuous glucose monitoring (CGM) to help target glucose control in extremely preterm infants who require intensive care. CGM however has not been used in babies who are being cooled. This study aims to determine if CGM can be safely used in these babies, and to use this alongside innovative methods to measure alternative fuels to optimise care of these vulnerable babies.

ELIGIBILITY:
Inclusion Criteria:

* Hypoxic ischaemic encephalopathy Informed parental consent

Exclusion Criteria:

* Known significant congenital malformation

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percent of time glucose levels measured on CGM are in target | From sensor insertion for up to the first 7 days of life
  Percent Time in target (2.6-10mmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Addenbrookes Hospital Trust, Cambridge, cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided